CLINICAL TRIAL: NCT00916123
Title: A Phase I Trial of Docetaxel/Prednisone Plus Fractionated 177Lu- J591 Anti-prostate-specific Membrane Antigen Monoclonal Antibody in Patients With Metastatic, Castrate-resistant Prostate Cancer
Brief Title: Docetaxel/Prednisone Plus Fractionated 177Lu- J591 Antibody for Metastatic, Castrate-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0812010139
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: castrate-resistant prostate cancer; CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 1 (Experimental): 177Lu-J591 at 20 mCi/dose
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: 177Lu-J591
- Dose Level 2 (Experimental): 177Lu-J591 at 25 mCi/dose
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: 177Lu-J591
- Dose Level 3 (Experimental): 177Lu-J591 at 30 mCi/dose
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: 177Lu-J591
- Dose Level 4 (Experimental): 177Lu-J591 at 35 mCi/dose
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: 177Lu-J591
- Dose Level 5 (Experimental): 177Lu-J591 at 40 mCi/dose
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: 177Lu-J591

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 by intravenous infusion over one hour on day 1 of a 21 day cycle.
  Other Names: Taxotere
Drug: Prednisone — 10 mg per day starting on cycle 1, day 1
  Other Names: Meticorten, Sterapred, Sterapred DS
Drug: 177Lu-J591 — Two infusions of 177Lu-DOTA-J591 at 20 mCi/dose will be given. The first infusion will be administered 2-3 days prior to docetaxel cycle 3. The second infusion will be administered two weeks later, i.e., day 13-15 of cycle 3.
  Arms: Dose Level 1
Drug: 177Lu-J591 — Two infusions of 177Lu-DOTA-J591 at 25 mCi/dose will be given. The first infusion will be administered 2-3 days prior to docetaxel cycle 3. The second infusion will be administered two weeks later, i.e., day 13-15 of cycle 3.
  Arms: Dose Level 2
Drug: 177Lu-J591 — Two infusions of 177Lu-DOTA-J591 at 30 mCi/dose will be given. The first infusion will be administered 2-3 days prior to docetaxel cycle 3. The second infusion will be administered two weeks later, i.e., day 13-15 of cycle 3.
  Arms: Dose Level 3
Drug: 177Lu-J591 — Two infusions of 177Lu-DOTA-J591 at 35 mCi/dose will be given. The first infusion will be administered 2-3 days prior to docetaxel cycle 3. The second infusion will be administered two weeks later, i.e., day 13-15 of cycle 3.
  Arms: Dose Level 4
Drug: 177Lu-J591 — Two infusions of 177Lu-DOTA-J591 at 40 mCi/dose will be given. The first infusion will be administered 2-3 days prior to docetaxel cycle 3. The second infusion will be administered two weeks later, i.e., day 13-15 of cycle 3.
  Arms: Dose Level 5

SUMMARY:
The purpose of this study is to test the effectiveness of the experimental drug, 177Lu-J591 antibody in combination with docetaxel chemotherapy against metastatic, castrate-resistant prostate cancer.

DETAILED DESCRIPTION:
This research is being done because the standard treatments for metastatic prostate cancer that is growing despite medical or surgical therapies are not curative. Existing treatments, such as the docetaxel used as part of this study, may work temporarily, but unfortunately the cancer continues to grow. This test drug, 177Lu-J591, is designed to seek out prostate cancer cells and deliver a lethal dose of radiation to the areas of cancer, but not to normal areas. Some of the normal organs (liver, kidney and bone marrow) do receive some radiation dose that is within the acceptable limits.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of prostate adenocarcinoma.
* Patient must have progressive metastatic prostate cancer despite adequate medical or surgical castration therapy.
* Serum testosterone < 50 mg/ml.
* Patients who have previously received docetaxel must meet BOTH of the the following criteria:

  * reason for docetaxel discontinuation must NOT have been progression of disease while receiving drug (i.e. progression of cancer must have been AFTER docetaxel discontinuation) AND
  * All docetaxel-related toxicities must have resolved to < grade 1 (with the exception of alopecia) and the pt must be eligible by other criteria

Exclusion Criteria:

* Use of red blood cell or platelet transfusions within 4 weeks of treatment.
* Use of hematopoietic growth factors within 4 weeks of treatment.-Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment.
* Bone scan demonstrating confluent lesions involving both axial and appendicular skeleton ("superscan").
* Prior radiation therapy encompassing >25% of skeleton.Prior treatment with 89Strontium or 153Samarium containing compounds (e.g. Metastron®, Quadramet®).
* Platelet count <150,000/mm3.
* Absolute neutrophil count (ANC) <2,000/mm3.
* Hematocrit <30 percent or Hemoglobin < 10 g/dL.
* Abnormal coagulation profile (PT or INR, PTT) > 1.3 x upper limit of normal (unless on therapeutic anticoagulation).
* -Serum creatinine >2.5 mg/dL.
* AST (SGOT) >2.5x ULN.
* Bilirubin (total) >1.5x ULN.
* Serum calcium >11 mg/dL.
* Active serious infection.
* Active angina pectoris or New York Heart Association Class III-IV.
* ECOG Performance Status >2.
* Life expectancy <6 months.
* Deep vein thrombosis and/or pulmonary embolus within 1 month of study entry.
* Other serious illness(es) which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.
* Prior anti-PSMA monoclonal antibody therapy with the exception of ProstaScint®.
* Prior investigational therapy within 6 weeks of treatment.
* Known history of HIV.
* Known history of myelodysplastic syndrome or leukemia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of fractionated 177Lu-DOTA-J591 administered concurrently with three-weekly docetaxel for the treatment of patients with metastatic, castrate-resistant prostate cancer. | 4 weeks post last J591 dose

SECONDARY OUTCOMES:
Determine the toxicity profile of concurrent docetaxel with fractionated 177Lu-DOTA-J591 | completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Batra JS, Niaz MJ, Whang YE, Sheikh A, Thomas C, Christos P, Vallabhajosula S, Jhanwar YS, Molina AM, Nanus DM, Osborne JR, Bander NH, Tagawa ST. Phase I trial of docetaxel plus lutetium-177-labeled anti-prostate-specific membrane antigen monoclonal antibody J591 (177Lu-J591) for metastatic castration-resistant prostate cancer. Urol Oncol. 2020 Nov;38(11):848.e9-848.e16. doi: 10.1016/j.urolonc.2020.05.028. Epub 2020 Jun 27. PMID 32600929